CLINICAL TRIAL: NCT05228691
Title: Long COVID: Evaluation of Physical and Functional Status
Brief Title: Prevalence of Long COVID-19 in the Canary Islands
Status: Recruiting | Type: Observational
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Principal Investigator, University of Las Palmas de Gran Canaria
Other Study IDs: COFC COVID
Record Dates: First submitted 2022-02-05; First posted 2022-02-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: physical therapy modality; Long COVID; post-acute COVID-19 syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long COVID: Participants will self-complete some questionnaires, while the rest of the variables will be evaluated by the evaluating physiotherapist.
  After the consultation, the evaluator himself will provide the participants with some recommendations that he should make. As support, a diptych has been made with different general activities to be developed by the participant. With the purpose of track this activity, they will be informed that they will be contacted once 6 months have passed since the evaluation (via phone call or SMS).
  Interventions: Other: Evaluation and Education

INTERVENTIONS:
Other: Evaluation and Education — A functional physical evaluation will be carried out and they will be informed about the characteristics of their symptoms. After the evaluation, they will be taught a guideline of exercises and recommendations.

SUMMARY:
With more than 246 million people diagnosed with coronavirus 2019 (COVID-19) around the world, many of whom have required medical attention for past 23 months, greater emphasis is being placed on post-acute care of COVID-19 survivors. According to recent data, millions of patients who have recovered from acute COVID-19 are experiencing persistent symptoms, which lead to disability and impaired activities of daily living.

Various terms have been used to describe the condition of patients who do not return to their initial health status to include post-acute sequelae of COVID-19, such as post-acute COVID syndrome (PACS) and Long COVID.

The growing global burden of COVID-19 suggests that the potential effects of Long COVID in public health are vast even if Long COVID is experienced by a small proportion of patients recovering from acute infection.

The ability to identify patients at high risk for Long COVID and forecasting medical resource requirements is of important clinical utility in the present.

In view of the large number of people surviving after infection with COVID-19 and that should require follow-up, determine which patients are at risk of have Long COVID and who require close monitoring is crucial. In this study, therefore, we set out to analyze what type of patient profile with COVID-19 who, after 12 weeks of having suffered the infection, experiences the signs and symptoms described by current literature.

DETAILED DESCRIPTION:
It is intended to develop a Cross-sectional Descriptive Observational Study. The investigation will be carried out following the guidelines of "Strengthening the Reporting of Observational Studies in Epidemiology" (STROBE).

A registry will be carried out at a multicenter level, in which a physical-functional evaluation will be carried out. of the patient who has suffered from COVID-19 and whose signs and symptoms last 12 weeks after its detection. This assessment is carried out by physiotherapists members of the entire Canarian Autonomous Community. Some quizzes will be completed with the assistance of a specific evaluator (physiotherapist), while that others will be self-completion.

In order to avoid bias and try to guarantee the highest methodological quality, prior to the recruitment, screening and evaluation of the participants, a specific training for all evaluators (physiotherapists). They will be addressed general theoretical content on COVID-persistent, justification and development logistics of the proposed study protocol, and implementation of the battery of evaluation tests.

The study participants will be recruited through non-recruited sampling probabilistic convenience.

The statistical analysis of the data will be carried out using the statistical software International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS) 27.

Categorical variables will be summarized using percentages and relative frequencies. The equality of proportions of the categories will be contrasted with the non-parametric tests Bi-nominal and Chi-Square (Goodness of fit). To test the possible association between categorical variables will use the Chi-square test or the exact test Fisher's.

To analyze the possible association between ordinal categorical variables, we will use to contrast Spearman's correlation coefficient. Numeric variables are summarized with the mean and standard deviation or by means of the median and the interquartile range, depending on whether or not the normality condition of the data is met.

To analyze the normality of the samples, the test of Kolmogorov-Smirnov or Shapiro-Wild. To compare the means of two independent samples, will use the Student's T test or the non-parametric U-Mann Whitney test, depending on whether or not the data normality condition.

In the case of means of 3 or more independent samples, will use the one-way ANOVA procedure or the non-parametric Kruskal Wallis test, depending on whether or not the normality condition of the data is met. To analyze the possible association between the numerical variables, the contrast of the coefficient of linear Pearson correlation.

According to the objectives and the associations that could be detected, it will be possible to use other statistical tools, or propose the construction of mathematical models predictive. The results will be considered statistically significant if p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have been positive for COVID-19 since the declaration of the state of alarm throughout the Spanish territory to deal with the health emergency situation caused by COVID-19 (March 14, 2020).
* Symptoms associated with COVID-19 at least after 12 weeks of its detection.
* Adequate cognitive and physical level to understand and perform the tests evaluation.

Exclusion Criteria:

* Present comorbidities prior to suffering from COVID-19 whose symptoms are resemble Post-acute COVID-19.
* Fibromyalgia.
* Chronic fatigue.
* Neuromuscular disease.
* Not having signed the informed consent.
* Person undergoing treatment for active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Autonomous Community of the Canary Islands presenting signs and symptoms related to COVID-19 and that last beyond 12 weeks from when disease debuted.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Post-COVID-19 Functional Status scale | 5 days before start the intervention
  The scale is ordinal, has 6 steps ranging from 0 (no symptoms) to 5 (death, D), and covers the full range of functional outcomes by focusing on limitations in usual tasks/activities, whether at home or at work/study, as well as lifestyle changes. The scale ratings are intuitive and can be easily understood by clinicians and patients alike.
Short Physical Performance Battery | Baseline at 0 minutes
  The Short Physical Performance Battery (SPPB) is a measure of physical performance that has been used to predict long-term disability and/or future institutionalization in adults aged 65 years and older. The test consists of three specific physical performance activities, scored from 0 to 4, with a summed score of 12. Higher scores reflect higher levels of function.
Aerobic capacity | Baseline at 0 minutes
  Aerobic capacity will be measured with the 1 minute sit to stand test: The purpose of the test is to assess the exercise capacity and leg muscle strength. The movement required is to get up from this chair with the legs straight and sit back continuing the repetitions as fast as possible within one minute.
  The mean number of 1-minute sit to stand test repetitions reported in the literature achieved ranged from 8.1 (patients with stroke) to 50.0 (young men).
Muscle Strength | Baseline at 0 minutes
  Muscle Strength will be measured with Medical Research Council (MRC) Scale : is a commonly used scale for assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction).
  This score was defined as the sum of the MRC scores of six muscles in the upper and lower limbs on both sides, so the score ranged from 60 (normal) to 0 (quadriplegic).
  The Criteria require that each of the six muscle groups be tested bilaterally, each scoring from 0 to 5.

SECONDARY OUTCOMES:
Musculoskeletal pain | 5 days before start the intervention
  Orebro Musculoskeletal Pain Questionnaire (OMPQ) This questionnaire is a clinical tool used to identify patients at risk of develop long-term chronic musculoskeletal problems. The questionnaire includes 21 questions, which are scored on a scale of 0 to 10, with a maximum possible score of 210 points.
Dyspnea | 5 days before start the intervention
  The Modified Medical Research Council (mMRC) Dyspnea Scale will be used. It´s a five-level rating scale based on the patient's perception of dyspnoea in daily activities.
  Grade 0: breathless with strenuous exercise; Grade 1: short of breath when hurrying on level ground or walking up a slight hill; Grade 2: walked slower than people of the same age on level ground, and experienced breathlessness or the need to stop to breathe when walking on level ground at their own pace; Grade 3: stop to breathe after walking about 100 yards, or after a few minutes on level ground; and Grade 4: too breathless to leave the house, or breathless when dressing or undressing.
Fatigue | 5 days before start the intervention
  The Fatigue Assessment Scale (FAS) is a tool that provides information about the physical and psychological aspects of fatigue, and provides a single overall score measuring its intensity.
  A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63
Physical activity | 5 days before start the intervention
  The International Physical Activity Questionnaires (IPAQ). This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in Metabolic Equivalent of Task (MET)-min/week and time spent sitting.
  A 7 items questionnaire, with open-ended questions surrounding individuals' last 7-day recall of physical activity.
Subjective health status assessment | 5 days before start the intervention
  Short Form-12 Health Survey (SF-12) is a generic short form health survey. It is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- University of Las Palmas de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carvalho-Schneider C, Laurent E, Lemaignen A, Beaufils E, Bourbao-Tournois C, Laribi S, Flament T, Ferreira-Maldent N, Bruyere F, Stefic K, Gaudy-Graffin C, Grammatico-Guillon L, Bernard L. Follow-up of adults with noncritical COVID-19 two months after symptom onset. Clin Microbiol Infect. 2021 Feb;27(2):258-263. doi: 10.1016/j.cmi.2020.09.052. Epub 2020 Oct 5. PMID 33031948
- [Result] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Result] Goertz YMJ, Van Herck M, Delbressine JM, Vaes AW, Meys R, Machado FVC, Houben-Wilke S, Burtin C, Posthuma R, Franssen FME, van Loon N, Hajian B, Spies Y, Vijlbrief H, van 't Hul AJ, Janssen DJA, Spruit MA. Persistent symptoms 3 months after a SARS-CoV-2 infection: the post-COVID-19 syndrome? ERJ Open Res. 2020 Oct 26;6(4):00542-2020. doi: 10.1183/23120541.00542-2020. eCollection 2020 Oct. PMID 33257910
- [Result] Iqbal FM, Lam K, Sounderajah V, Clarke JM, Ashrafian H, Darzi A. Characteristics and predictors of acute and chronic post-COVID syndrome: A systematic review and meta-analysis. EClinicalMedicine. 2021 May 24;36:100899. doi: 10.1016/j.eclinm.2021.100899. eCollection 2021 Jun. PMID 34036253